CLINICAL TRIAL: NCT03147261
Title: Impacto de Una intervención Integral Sobre el Riesgo cardiometabólico en niños Con Obesidad Central: Estudio de Marcadores genéticos y epigenéticos
Brief Title: Impact of Comprehensive Intervention on the Cardiometabolic Risk in Children With Central Obesity (IGENOI)Obesity
Acronym: IGENOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNavarre
Record Dates: First submitted 2017-05-03; First posted 2017-05-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- lifestyle intervention (Experimental): Intensive follow up in lifestyle factors with a reduced calorie DM , physical activity and behavioural therapy.
  Interventions: Other: Lifestyle intervention
- No intervention (No Intervention): Healthy diet recommendations following the usual pediatric advice

INTERVENTIONS:
Other: Lifestyle intervention — Intensive changes in lifestyle with a reduced calorie mediterranean diet, physical activity and behavioral therapy
  Other Names: No intervention
  Arms: lifestyle intervention

SUMMARY:
Central obesity, present in the metabolic syndrome (MS), is associated with increased risk of insulin resistance (RI). The aim of the project is to evaluate the protective effect of comprehensive intervention (Mediterranean diet + physical activity) in the development of RI in children with central obesity based on genetic and epigenetic markers.

DETAILED DESCRIPTION:
Objectives: 1) Apply a comprehensive therapeutic nutrition intervention program for monitoring the Mediterranean Diet (DM) slightly hypocaloric along with increased physical activity in children with central obesity 7-16 years). 2) Measure the effectiveness of this program by assessing changes in body composition, lifestyle and biological and molecular parameters (genetic and epigenetic).

Methodology: test randomized, longitudinal, controlled, two-year intervention field comparing a sample of 120 subjects from 7 to 16 years with central obesity, the effect of two interventions: a) intensive on lifestyle with a reduced calorie DM , physical activity and behavioral therapy, b) non-intensive with healthy diet recommendations following the usual pediatric advice. At 2, 6, 12 and 24 months after follow up changes will be assessed: a) the HOMA index, body fat, and the cardiovascular risk factors, b) diet, sleep patterns, physical exercise using questionnaires and accelerometers (intervention group), and c) the quality of life. genetic and epigenetic markers will be evaluated by genotyping SNPs genes related to RI; and the analysis of: a) DNA methylation in genes related to insulin resistance, b) expression of microRNAs and target genes related to insulin resistance and c) measure the length of telomeres. The therapeutic program will consist of individual sessions and group workshops for the patient and the family.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the child, parent or guardian. 3. waist circumference above the 90th percentile 4. Motivation and willingness to be assigned to either group, and do their utmost to follow protocol assigned.

5. Possibility of involvement in days of intensive phase (week 0, 1, 2, 3, 4, 5, 6, 7 and 8) and once a month until 6 months later at 4 months and every 6 months during the second year.

Exclusion Criteria:

1. Pre-Diabetes
2. Presence of other diseases
3. Pharmacotherapy
4. Monitoring special diets
5. Food intolerance
6. Regular alcohol consumption
7. Drug
8. Psychiatric illness or eating disorder
9. People without telephone or Internet access

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-12; Primary Completion 2018-02 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
changes in the HOMA index | At 2, 6, 12 and 24 months after follow up
  changes will be assessed in the HOMA index

SECONDARY OUTCOMES:
genetic and epigenetic markers will be evaluated | At 2, 6, 12 and 24 months after follow up
  genetic and epigenetic markers will be evaluated by genotyping SNPs genes related to RI; and the analysis of: a) DNA methylation in genes related to insulin resistance, b) expression of microRNAs and target genes related to insulin resistance and c) measure the length of telomeres

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Marti, PhD, Study Director — University of Navarra
Locations (1):
- UNavarre, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morell-Azanza L, Ojeda-Rodriguez A, Azcona-SanJulian MC, Zalba G, Marti A. Associations of telomere length with anthropometric and glucose changes after a lifestyle intervention in abdominal obese children. Nutr Metab Cardiovasc Dis. 2020 Apr 12;30(4):694-700. doi: 10.1016/j.numecd.2019.12.002. Epub 2019 Dec 10. PMID 32007334
- [Derived] Morell-Azanza L, Ojeda-Rodriguez A, Ochotorena-Elicegui A, Martin-Calvo N, Chueca M, Marti A, Azcona-San Julian C. Changes in objectively measured physical activity after a multidisciplinary lifestyle intervention in children with abdominal obesity: a randomized control trial. BMC Pediatr. 2019 Apr 4;19(1):90. doi: 10.1186/s12887-019-1468-9. PMID 30947686